CLINICAL TRIAL: NCT05216588
Title: Pre-exposure Prophylaxis of SARS-CoV-2 Infection (COVID-19) by Monoclonal Antibodies with Early Access Authorization in Immunocompromised Patients. a Prospective Cohort.
Acronym: PRECOVIM
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS0166s PRECOVIM; 2021-006961-39 (EudraCT Number)
Record Dates: First submitted 2022-01-25; First posted 2022-01-31 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: COVID-19; Immunocompromised Host
Keywords: Post-Exposure Prophylaxis; Antibodies Monoclonal; Neutralizing Antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, nasopharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- EVUSHELD (tixagévimab/cilgavimab) 300 mg: Patients who may be included in this group are patients eligible for prophylaxis treatments for COVID-19, under a cohort Temporary Authorization for Use (ATUc) of EVUSHELD 300mg. Patient are treated and monitored according to the Therapeutic Use Protocols specific for EVUSHELD defined by the ANSM.
  In addition to their follow-up planned for usual care (including protocol for ATU), they are invited to participate in the research.
- EVUSHELD (tixagévimab/cilgavimab) 600 mg: Patients who may be included in this group are patients eligible for prophylaxis treatments for COVID-19, under a cohort Temporary Authorization for Use (ATUc) of EVUSHELD 600mg. Patient are treated and monitored according to the Therapeutic Use Protocols specific for EVUSHELD defined by the ANSM.
  In addition to their follow-up planned for usual care (including protocol for ATU), they are invited to participate in the research.

SUMMARY:
This prospective cohort of patients, receiving pre exposure prophylaxis by Anti-SARS-CoV-2 Monoclonal Antibodies, is designed to evaluate the treatment protection against SARS-CoV-2 variants of concerns

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years-old or more)
* Patient who received the first administration of Evusheld at 300 mg for less than 4 months and should receive a second dose, according to French recommendations OR Patient scheduled to receive or having received less than a month ago an injection of anti-SARS-CoV-2 monoclonal antibodies, as pre-exposure prophylaxis at 600 mg, according to the French SARS-CoV-2 RT recommendations
* qPCR negative at baseline
* SARS-CoV-2 RT-qPCR Negative at inclusion
* Patients who remain seronegative after a complete COVID-19 vaccination schedule
* Immunocompromised patients :

Hemopathy : chronic lymphoid leukemia, non hodgkin's lymphoma, HSCT Transplant recipient : kidney, liver, lungs Patients receiving anti CD20 or others immunosuppressor

* Life expectancy > 3 months
* Social security affiliation
* Lack of a legal protection measure
* Signed informed consent

Exclusion Criteria:

* Participation to another clinical study
* State medical aid
* Ongoing or scheduled plasmapheresis or immunoadsorption
* Pregnant / lactating woman
* Patient whose isolation period is underway following contact with a confirmed case of SARS-CoV2 infection
* Hypersensitivity to one of the active substances or to one of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who may be included in the cohort are patients eligible for prophylaxis treatments for COVID-19, under a cohort Temporary Authorization for Use (ATUc) or full market approval. In case of ATUc, patient are treated and monitored according to the Therapeutic Use Protocols specific for each ATU treatment defined by the ANSM.
  In addition to their follow-up planned for usual care (including protocol for ATU), they are invited to participate in the research.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Neutralizing antibody activity | Month 1
Neutralizing antibody activity | Month 2
Neutralizing antibody activity | Month 3
Neutralizing antibody activity | Month 4
Neutralizing antibody activity | Month 5
Neutralizing antibody activity | Month 6
Neutralizing antibody activity | Month 9
Neutralizing antibody activity | Month 12

SECONDARY OUTCOMES:
Proportion of subjects who have a positive SARS-CoV-2 RT-qPCR) and symptoms of SARS-CoV-2 infection | Month 12
Proportion of subjects hospitalized related to a RT-qPCR confirmed SARS-CoV-2 infection during prophylaxis period | Month 12
Proportion of patients infected with a resistant variant | Month 12
Proportion of patients with treatment AE | Month 12
Severity of treatment AE | Month 12
Proportion of patients with SAE | Month 12
Proportion of patients with suspended prophylaxis due to adverse event | Month 12
Variability of the individual pharmacokinetic parameters of the two monoclonal antibodies and covariates influencing it | Month 1
Variability of the individual pharmacokinetic parameters of the two monoclonal antibodies and covariates influencing it | Month 2
Variability of the individual pharmacokinetic parameters of the two monoclonal antibodies and covariates influencing it | Month 3
Variability of the individual pharmacokinetic parameters of the two monoclonal antibodies and covariates influencing it | Month 4
Variability of the individual pharmacokinetic parameters of the two monoclonal antibodies and covariates influencing it | Month 5
Variability of the individual pharmacokinetic parameters of the two monoclonal antibodies and covariates influencing it | Month 6
Variability of the individual pharmacokinetic parameters of the two monoclonal antibodies and covariates influencing it | Month 9
Variability of the individual pharmacokinetic parameters of the two monoclonal antibodies and covariates influencing it | Month 12
Relations between the concentrations of the two monoclonal antibodies and the levels of anti-S and anti-N antibodies | Month 1
Relations between the concentrations of the two monoclonal antibodies and the levels of anti-S and anti-N antibodies | Month 2
Relations between the concentrations of the two monoclonal antibodies and the levels of anti-S and anti-N antibodies | Month 3
Relations between the concentrations of the two monoclonal antibodies and the levels of anti-S and anti-N antibodies | Month 4
Relations between the concentrations of the two monoclonal antibodies and the levels of anti-S and anti-N antibodies | Month 5
Relations between the concentrations of the two monoclonal antibodies and the levels of anti-S and anti-N antibodies | Month 6
Relations between the concentrations of the two monoclonal antibodies and the levels of anti-S and anti-N antibodies | Month 9
Relations between the concentrations of the two monoclonal antibodies and the levels of anti-S and anti-N antibodies | Month 12
Relations between the concentrations of the two monoclonal antibodies and the neutralizing activity of the serum towards the omicron variant of SARS-CoV-2 | Month 1
Relations between the concentrations of the two monoclonal antibodies and the neutralizing activity of the serum towards the omicron variant of SARS-CoV-2 | Month 2
Relations between the concentrations of the two monoclonal antibodies and the neutralizing activity of the serum towards the omicron variant of SARS-CoV-2 | Month 3
Relations between the concentrations of the two monoclonal antibodies and the neutralizing activity of the serum towards the omicron variant of SARS-CoV-2 | Month 4
Relations between the concentrations of the two monoclonal antibodies and the neutralizing activity of the serum towards the omicron variant of SARS-CoV-2 | Month 5
Relations between the concentrations of the two monoclonal antibodies and the neutralizing activity of the serum towards the omicron variant of SARS-CoV-2 | Month 6
Relations between the concentrations of the two monoclonal antibodies and the neutralizing activity of the serum towards the omicron variant of SARS-CoV-2 | Month 9
Relations between the concentrations of the two monoclonal antibodies and the neutralizing activity of the serum towards the omicron variant of SARS-CoV-2 | Month 12
Relations between the concentrations of the two monoclonal antibodies and the risk of infection by the omicron variant of SARS-CoV-2 | Month 1
Relations between the concentrations of the two monoclonal antibodies and the risk of infection by the omicron variant of SARS-CoV-2 | Month 2
Relations between the concentrations of the two monoclonal antibodies and the risk of infection by the omicron variant of SARS-CoV-2 | Month 3
Relations between the concentrations of the two monoclonal antibodies and the risk of infection by the omicron variant of SARS-CoV-2 | Month 4
Relations between the concentrations of the two monoclonal antibodies and the risk of infection by the omicron variant of SARS-CoV-2 | Month 5
Relations between the concentrations of the two monoclonal antibodies and the risk of infection by the omicron variant of SARS-CoV-2 | Month 6
Relations between the concentrations of the two monoclonal antibodies and the risk of infection by the omicron variant of SARS-CoV-2 | Month 9
Relations between the concentrations of the two monoclonal antibodies and the risk of infection by the omicron variant of SARS-CoV-2 | Month 12
Relationship between the concentrations of the two monoclonal antibodies and the risk of of adverse effects. | Month 1
Relationship between the concentrations of the two monoclonal antibodies and the risk of of adverse effects. | Month 2
Relationship between the concentrations of the two monoclonal antibodies and the risk of of adverse effects. | Month 3
Relationship between the concentrations of the two monoclonal antibodies and the risk of of adverse effects. | Month 4
Relationship between the concentrations of the two monoclonal antibodies and the risk of of adverse effects. | Month 5
Relationship between the concentrations of the two monoclonal antibodies and the risk of of adverse effects. | Month 6
Relationship between the concentrations of the two monoclonal antibodies and the risk of of adverse effects. | Month 9
Relationship between the concentrations of the two monoclonal antibodies and the risk of of adverse effects. | Month 12
Anti-S et Anti- N antibodies levels | Month 1
Anti-S et Anti- N antibodies levels | Month 2
Anti-S et Anti- N antibodies levels | Month 3
Anti-S et Anti- N antibodies levels | Month 4
Anti-S et Anti- N antibodies levels | Month 5
Anti-S et Anti- N antibodies levels | Month 6
Anti-S et Anti- N antibodies levels | Month 9
Anti-S et Anti- N antibodies levels | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LEVY, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Lamballerie X, Martin-Blondel G, Dupont A, Izopet J, Mentre F, Kamar N, Autran B, Paintaud G, Caillard S, le Bourgeois A, Richez C, Couzi L, Xhaard A, Marjanovic Z, Avouac J, Jacquet C, Anglicheau D, Cheminant M, Yazdanpanah Y, Guyen SN, Terrier B, Gottenberg JE, Besson C, Letrou S, Kali S, Angoulvant D, Sanchez VP, Tardivon C, Blancho G, Levy V. Low serum neutralization of Omicron variants a month after AZD7442 prophylaxis initiation. J Infect. 2023 Jan;86(1):66-117. doi: 10.1016/j.jinf.2022.10.006. Epub 2022 Oct 8. No abstract available. PMID 36216187